CLINICAL TRIAL: NCT03842072
Title: The Collar Post Anterior Cervical Spine Surgery (C-PASS) Study: Project Proposal for a Multi-Center Randomized Trial Evaluating the Impact of Post-Operative Bracing on Clinical Outcomes After Anterior Cervical Discectomy and Fusion.
Brief Title: The Collar Post Anterior Cervical Spine Surgery Study
Acronym: C-PASS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-PASS
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Cervical Radiculopathy; Cervical Myelopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No post-operative bracing (No Intervention): patients in this arm will not be prescribed a cervical collar following anterior cervical discectomy and fusion surgery
- Post-operative bracing (Active Comparator): Patients in this arm will be prescribed a cervical collar following anterior cervical discectomy and fusion surgery.
  Interventions: Device: Cervical collar

INTERVENTIONS:
Device: Cervical collar — cervical collars prescribed will be use immediately following anterior cervical discectomy and fusion surgery.
  Arms: Post-operative bracing

SUMMARY:
The Anterior Cervical Discectomy and Fusion (ACDF) represents one of the most commonly performed spinal operations internationally, often in the context of symptomatic radiculopathy or myelopathy secondary to cervical degenerative disease. Approximately half of surgeons continue to prescribe a period of post-operative bracing with a cervical collar. However, there is currently no high quality evidence available to support the routine use of post-operative bracing after ACDF; further, braces are expensive and have been associated with a variety of local complications. In summary, the current lack of evidence, and lack of consensus amongst surgeons, regarding best practices in the use of post-operative bracing after ACDF, places the surgeon and the patient in a precarious position.

Our randomized trial comparing the impact of 6 weeks of post-operative bracing with a rigid cervical collar vs. no post-operative bracing, on a variety of clinical and radiological outcomes, for adult patients with cervical radiculopathy and/or myelopathy undergoing single or multi-level ACDF.

DETAILED DESCRIPTION:
The Anterior Cervical Discectomy and Fusion (ACDF) represents one of the most commonly performed spinal operations internationally, often in the context of symptomatic radiculopathy or myelopathy secondary to cervical degenerative disease. Approximately half of surgeons continue to prescribe a period of post-operative bracing with a cervical collar. However, there is currently no high quality evidence available to support the routine use of post-operative bracing after ACDF; further, braces are expensive and have been associated with a variety of local complications. In summary, the current lack of evidence, and lack of consensus amongst surgeons, regarding best practices in the use of post-operative bracing after ACDF, places the surgeon and the patient in a precarious position.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 18 and 80;
2. presenting with cervical radiculopathy and/or myelopathy to one of the study centers;
3. deemed appropriate by the attending surgeon involved for a one, two or three level plated ACDF or a one-level ACDF with a standalone interbody cage; and
4. able to cooperate in the completion of all study consents, forms and documents. 5. Participants who are able to speak, read and write at an elementary school level

Exclusion Criteria:

1. those with previous cervical surgery;
2. those undergoing single or multi-level plated ACDF for a diagnosis related to malignancy, infection or trauma;
3. those undergoing a single or multi-level plated ACDF augmented with a posterior cervical fusion or posterior cervical decompression and fusion;
4. those undergoing a multi-level non-plated ACDF;
5. those undergoing ACDF at greater than three levels, and;
6. those with a pre-existent neurological or mental disorder which would preclude accurate evaluation and follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Neck Disability index | 6 month
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life.

SECONDARY OUTCOMES:
Neck Disability Index | 3 and 12 month
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life.
EQ-5D | 3, 6, 12 month
  a standardized instrument for measuring generic health status.
Visual analog score | 3, 6, 12 month
  a measurement instrument for pain where pain is measured from a score of 0 (represents no pain), and 10 (most pain, or worst pain imaginable.
Plain Xray Radiography | 6 week, 12 month
  An X-ray is a quick, painless test that produces images of the structures inside your body

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson Wilson, MD, FRCSC, Principal Investigator — Unity Health Toronto
Locations (2):
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - Hôpital Général de Montréal Montreal General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No